CLINICAL TRIAL: NCT00782093
Title: A Phase 1 Ascending and Parallel Group Trial to Establish the Safety, Tolerability and Pharmacokinetics Profile of Volociximab (Alpha 5 Beta 1 Integrin Antagonist) in Subjects With Neovascular Age- Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ophthotech Corporation (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M200
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2012-06

CONDITIONS: Age-related Macular Degeneration
Keywords: AMD
MeSH Terms: conditions — Macular Degeneration | interventions — volociximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: volociximab — volociximab intravitreal injection

SUMMARY:
The objectives of this study are to evaluate the safety, tolerability, and pharmacokinetic profile of volociximab intravitreous injection in subjects with subfoveal choroidal neovascularization secondary to age-related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Subfoveal choroidal neovascularization (CNV) due to AMD (i.e., predominantly classic, minimally classic or occult no classic) as documented by fluorescein angiogram.

Exclusion Criteria:

* Any prior treatment for AMD or any intravitreal treatment for any indication in the study eye prior to the screening visit, except oral supplements of vitamins and minerals.
* Previous or concomitant therapy with intravitreous corticosteroids.
* Any of the following underlying diseases including:
* Diabetic retinopathy
* History or evidence of severe cardiac disease (e.g., NYHA Functional Class III or IV - see Appendix 19.6), history or clinical evidence of unstable angina, acute coronary syndrome, myocardial infarction or revascularization within last 6 months, ventricular tachyarrythmias requiring ongoing treatment.
* History or evidence of clinically significant peripheral vascular disease, such as intermittent claudication or prior amputation.
* Clinically significant impaired renal (serum creatinine >2.5 mg/dl or s/p renal transplant or receiving dialysis) or hepatic function. Patients with results outside these ranges may be enrolled in consultation with Ophthotech.
* Stroke (within 12 months of trial entry).
* Any major surgical procedure within one month of trial entry.
* Previous therapeutic radiation in the region of the study eye.
* Any treatment with an investigational agent in the past 60 days for any condition.
* Women who are pregnant or nursing.
* Known serious allergies to the fluorescein dye used in angiography, to the components of the ranibizumab formulation, or to the components of the volociximab formulation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The primary safety endpoint is the presence of any dose limiting toxicity (DLT) | 2 years